CLINICAL TRIAL: NCT06887452
Title: Pharmacist-Led Treat-to-Target Urate Lowering Therapy in Patients in Gout (Pharm-UP) Study
Brief Title: Pharmacist-Led Treat-to-Target Urate Lowering Therapy in Patients With Gout
Acronym: Pham-UP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMMA-005-24F; CX002995 (Other Grant/Funding Number: VA CSR&D)
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Gout; Gouty Arthritis
MeSH Terms: conditions — Gout; Arthritis, Gouty

STUDY DESIGN:
Intervention Model Description: Randomized multicenter, parallel-group study that will compare a pharmacist-led / telehealth delivered intervention to usual care in gout management
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pharmacist-Led (Experimental): Veterans will participate in regular telehealth visits with study pharmacists. Serum urate lab tests will be ordered during dose escalation phase of gout treatment.
  Interventions: Other: Pharmacist-Led
- Usual care (No Intervention): Veterans will receive standard care from their primary care provider for the management of their gout.

INTERVENTIONS:
Other: Pharmacist-Led — Pharmacist will conduct regular telehealth visits with Veterans during dose escalation phase of gout treatment
  Arms: Pharmacist-Led

SUMMARY:
This study will compare two different approaches to manage medications that lower uric acid levels. This study will be conducted at five VA medical centers across the United States and will take 4-5 years to complete. Individual participation will last up to two years.

DETAILED DESCRIPTION:
This project will quantify and compare the effects of a pharmacist-led telehealth-delivered intervention versus usual care on arthritis flare burden and serum urate goal achievement in 310 U.S. Veterans with gout enrolled from five VA medical centers. The project will quantify the effects of the intervention on patient-reported outcomes (improvements in health-related quality of life, pain interference, and participant global assessment).

ELIGIBILITY:
Inclusion Criteria:

* US Veterans over the age of 18 years with physician-diagnosed
* Documented hyperuricemia (SU >6.8 mg/dL)
* Satisfy ACR/EULAR gout classification criteria
* Report 1 or more flares in the prior 6 months
* Receipt of a new ULT prescription (allopurinol or febuxostat) initiated by a primary care provider or longer term ULT but otherwise satisfy the flare/SU criteria

Exclusion Criteria:

* Any patient intolerant or unable to take ULTs (allopurinol or febuxostat)
* Patients with a rheumatology encounter within the prior 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
flare occurrence | during year two
  The occurrence of two or more flares during year 2.
serum urate at goal | at end of year one
  Achievement of serum urate <6 mg/dL at end of year one.

SECONDARY OUTCOMES:
Veterans RAND 12 (VR-12) | Baseline visit, Months 6, 12, 18, and 24
  Quality of life instrument to assess components of physical and mental health. The survey asks about a patient's views on their health. The information will keep track of how a patient feels and how well they are able to do their usual activities. Scores include ranking their health from excellent to poor, whether physical or emotional health or pain limits activities or accomplishments, whether their health interferes with social activities and lastly asks patients to compare their physical and emotional health to one year ago. The scales range from not-at-all through all the time.
Patient Reported Outcomes Measurement Information System (PROMIS) | Baseline visit, Months 6, 12, 18, and 24
  Survey to assess pain on relevant aspects of a patient's life within the last 7 days. The survey asks whether or not pain interfered with enjoyment, concentration, outside-of-home tasks, and socialization. The scale is at a not at all (1) through very much (5).
Gout-related patient global assessment | Baseline visit, Months 6, 12, 18, and 24
  Participants will complete a rating scale on all the ways gout affects them on a 0-100 scale ranging from very well to very poor.

CONTACTS AND LOCATIONS:
Overall Officials: Ted R. Mikuls, Principal Investigator — Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE
Locations (5):
- United States (5):
  - Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No